CLINICAL TRIAL: NCT03268486
Title: Evaluation of a Novel Signal Acquisition Technique for Intrapartum Cardiotocography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Ana Catarina Reis de Carvalho, Resident, University of Lisbon
Other Study IDs: ULisbon TAECG
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Labor Fetal Anoxia; Fetal Monitoring
Keywords: Fetal monitoring; cardiotocography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple monitoring: Pregnant women with singleton term pregnancies, spontaneous or induced/augmented labor, cephalic presentation, > 18 years of age, able to provide written informed consent, no contraindications to internal FHR monitoring and no known contraindication to vaginal delivery. After giving written informed consent, women will be simultaneously monitored with scalp electrode, Doppler, trans-abdominal ECG, abdominal EHG and TOCO, as soon as internal monitoring is possible.

SUMMARY:
Cardiotocography (CTG) is widely used during labour wards in industrialised countries and consists of fetal heart rate and uterine contraction monitoring. The main aim is to identify fetuses that are being poorly oxygenated during labour and require medical intervention to revert the situation or expedite delivery.

The need for technical development of CTG is well-recognized, as some of the existing techniques are prone to signal loss and contamination from the maternal heart rate, while others are invasive and have established contra-indications. They also limit maternal mobilisation, contributing to maternal dissatisfaction, and possibly to adverse maternal and neonatal outcomes.

New techniques for CTG acquisition will shortly be made available by a leading technological company, providing non-invasive monitoring and allowing full maternal mobilisation, and with the potential to change the way labour is conducted in high-resource countries. There is a need for a systematic evaluation of their clinical performance and benefit.

DETAILED DESCRIPTION:
First phase of the study will start in October 2017 in labor wards at Hospital de Santa Maria, Lisbon where performing continuous cardiotocographic fetal monitoring with conventional Doppler technology is the routine procedure. Through a collaboration with Phillips (Boeblingen, Germany) we will have access to a transabdominal ECG/EHG recorder that has high accuracy/reliability and Bluetooth technology providing mobility and and more comfort for mothers. This new device works through five disposable electrodes that are positioned on the maternal abdomen in a standardized manner: one electrode is placed near the umbilicus, a second is placed above the symphysis pubis in a vertical line from the umbilicus, a third and a fourth are placed on opposite sides of the abdomen horizontal to the umbilicus; the ground is placed on the upper right side. Women will be informed of the study by posters and leaflets distributed during the antenatal period and on arrival at labor wards. The inclusion criteria are singleton term pregnancies, spontaneous or induced/augmented labor, cephalic presentation, > 18 years of age, able to provide written informed consent, no contraindications to internal FHR monitoring and no known contraindication to vaginal delivery. Patients with risk factors for intrapartum hypoxia will also be included. After giving written informed consent, women will be simultaneously monitored with scalp electrode, Doppler, trans-abdominal ECG, abdominal EHG and TOCO, as soon as internal monitoring is possible. The maternal abdominal skin will be prepared for low impedance by gentle excoriation of the surface skin cells. Monitoring will be maintained until as close to delivery as possible, and the three FHR signals will be conveyed to a computer acquisition storage system for offline analysis. We aim a sample size of 100 participants. EHG and TOCO will be compared for signal loss, contraction frequency, and contraction area. Transabdominal ECG and Doppler will be compared in terms of signal loss, and with internal ECG regarding signal accuracy. The signal quality will be analysed separately for each monitoring method for the time during which the FHR recorded. As the two FHR modalities do not share a common time clock, synchronisation should be achieved by cross correlating the two heart rate files and locating the peak correlation. The clinical management of labour will be uniquely on the basis of external Doppler ultrasound CTG recordings. Both signals will also be compared for coincidences with MHR determined by maternal ECG with FHR determined by internal ECG. The abdominal fECG monitor calculates the MHR as well as the FHR simultaneously. It uses the height and the width of the QRS complex, both of which are linked to the size of the heart, to differentiate between the fetal and maternal heart signals. Women will be encouraged to perform a sequence of standardized exercises, in the presence of the investigator, and the periods when the mother is lying down, sitting, standing and walking will be recorded.

A subgroup analysis will be performed in the different stages of labour, particularly during maternal pushing, as well as in women with different skin colour and body mass index categories and in the different positions they adopt. Both umbilical cord arterial and venous blood sampling will be performed for the diagnosis of newborn metabolic acidosis, as soon as possible after birth. Data on basic demographic characteristics, pregnancy complications, course of labor, and neonatal outcome will be obtained.

In the second phase of the study, we want to know if the different traces acquired from the same fetus through transabdominal ECG and Doppler CTG may have different interpretations and may lead to different obstetric attitudes. In order to do that we will retrospectively analyze all the independent traces through a computer analysis (Omniview-SisPorto program). This system emits visual and sound alerts when features associated with poor fetal oxygenation are detected and has been shown to provide analysis that is in good agreement with a consensus of experts. The main outcome will be the agreement of alerts displayed by each signal acquisition technique regarding the same fetus.

ELIGIBILITY:
Inclusion Criteria:

* Singleton term pregnancies, spontaneous or induced/augmented labor, cephalic presentation, > 18 years of age, able to provide written informed consent, no contraindications to internal FHR monitoring and no known contraindication to vaginal delivery. Patients with risk factors for intrapartum hypoxia will also be included.

Exclusion Criteria:

* Do not give a written consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women (pregnant)
Study Population: All pregnant women in labour at Hospital de Santa Maria, Lisbon
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Signal quality | The analysis will be made at the end of the recruiting phase (that will have 3 months of duration)
  Transabdominal ECG and Doppler will be compared in terms of signal loss, and with internal ECG regarding signal accuracy. The signal quality will be analysed separately for each monitoring method for the time during which the FHR recorded.

IPD SHARING:
Plan to Share IPD: No